CLINICAL TRIAL: NCT01820468
Title: Adapting a Critical Time Intervention Model for Veterans on a Psychiatric Inpatient Unit
Brief Title: Adapting a Model for Veterans on a Psychiatric Inpatient Unit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated before any participants were enrolled due to unforseen problems with participant enrollment and study design.
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01715
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-12

CONDITIONS: Conditions: Serious Mental Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adapted critical time intervention team (Experimental): Community-based team will help facilitate early inpatient discharge and re-entry into the community.
  Interventions: Behavioral: Adapted critical time intervention team
- Regular inpatient care (No Intervention)

INTERVENTIONS:
Behavioral: Adapted critical time intervention team
  Arms: Adapted critical time intervention team

SUMMARY:
This randomized controlled study tests an adapted critical time intervention model for veterans discharged from a psychiatric inpatient unit. It is hypothesized that veterans on the inpatient unit who are assigned to such a community-based team will have shorter lengths of inpatient stay and better mental health. There have been few developments of community-based models of care in the post-deinstitutionalization era of short inpatient stays and the results of the study may inform how inpatient stays can be further reduced.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the psychiatric inpatient unit for at least 4 days
2. Willing to participate in community-based treatment

Exclusion Criteria:

1. Actively suicidal or homicidal
2. Dementia
3. Drug or alcohol detoxification
4. Physician emergency certificate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Length of inpatient stay | 1 month follow-up

SECONDARY OUTCOMES:
Mental health functioning | 1 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jack Tsai, Ph.D., Principal Investigator — VA Connecticut Healthcare System